CLINICAL TRIAL: NCT04617314
Title: A Phase I Study to Evaluate the Safety, Pharmacokinetics, and Effect of RC108-ADC For Injection in Subjects With c-Met Positive Advanced Malignant Solid Tumors
Brief Title: A Study of RC108-ADC in Subjects With Advanced Malignant Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: RemeGen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC108-C001
Record Dates: First submitted 2020-10-30; First posted 2020-11-05 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-03

CONDITIONS: Solid Tumor
Keywords: c-Met positive; solid tumor
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RC108 (Experimental): Participants will be allocated to one of the following dose groups: 0.1, 0.3, 0.9, 1.5, 2.0, 2.5, and 3.0mg/kg, and receive a treatment of RC108-ADC followed by 21 days of dose limited toxicity (DLT) observation period.
  Interventions: Drug: RC108

INTERVENTIONS:
Drug: RC108 — RC108 for injection is a novel antibody-drug conjugate, with a c-Met-targeting antibody and a microtube inhibitor.
  Other Names: RC108 for injection

SUMMARY:
This study will evaluate the safety, pharmacokinetics, and effect of RC108-ADC for injeciton in subjects with c-Met positive advanced malignant solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary agreement to provide written informed consent.
2. Male or female, aged between 18 to 70 years.
3. Predicted survival for ≥ 12 weeks.
4. Diagnosed with histologically or cytologically confirmed locally advanced or metastatic solid tumors.
5. Measurable lesion according to RECIST 1.1.
6. c-Met positive as confirmed by the central laboratory. The subject is able to provide specimens from primary or metastatic lesions for c-Met tests.
7. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.
8. Adequate organ function, evidenced by the following laboratory results within 7 days prior to the study treatment:
9. Cardiac ejection fraction ≥ 50%. Median QTc < 450 ms. Hemoglobin ≥ 9g/dL; Absolute neutrophil count ≥ 1.5×10^9 /L Platelets ≥ 100×10^9 /L; Total bilirubin ≤ 1.5× ULN; AST and ALT ≤ 2.5×ULN and ≤ 5 x ULN with hepatic metastasis; Serum creatinine ≤1.5×ULN.
10. All female subjects will be considered to be of child-bearing potential unless they are postmenopausal, or have been sterilized surgically. Female subjects of child-bearing potential must agree to use two forms of highly effective contraception. Male subjects and their female partner who are of child-bearing potential must agree to use two forms of highly effective contraception.
11. Willing to adhere to the study visit schedule and the prohibitions and restrictions specified in this protocol.

Exclusion Criteria:

1. Known hypersensitivity to the components of RC108-ADC.
2. Toxicity of previous anti-tumor treatment not recovered to CTCAE (v5.0) Grade 0-1 (with exception of Grade 2 alopecia).
3. Uncontrolled pericardial effusion or cardiac tamponade, or pleural or abdominal effusion with clinical symptoms.
4. History of receiving any anti-cancer drug/biologic treatment within 4 weeks prior to trial treatment.
5. History of major surgery within 4 weeks of planned start of trial treatment.
6. Has received a live virus vaccine within 4 weeks of planned start of trial treatment.
7. Currently known active infection with HIV or tuberculosis.
8. Diagnosed with HBsAg, HBcAb positive and HBV DNA copy positive, or HCVAb positive.
9. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
10. History of other malignancy within the previous 5 years, except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, or cancers with a similar curative outcome as those mentioned above.
11. Known central nervous system metastases.
12. Uncontrolled hypertension, diabetes, pulmonary fibrosis, acute lung disease, Interstitial lung disease, or liver cirrhosis;
13. Pregnancy or lactation.
14. Assessed by the investigator to be unable or unwilling to comply with the requirements of the protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | From the day of ICF signment to 28 days after the day of the last treatment
  Adverse events was assessed by investigator(s) according to NCI-CTCAE v4.03
Maximum Tolerated dose of RC108 | 21 days after first treatment.
  The dose level in which >= 2 out of 6 patients have dose-limiting toxicity (DLT). The MTD is defined as the previous dose level.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 24 months
  Objective Response Rate was defined as the percentage of participants with a complete response (CR) or partial response (PR)
Progression Free Survival (PFS) | 24 months
  Progression-free Survival (PFS) (median) was determined using the number of months measured from the initial date of treatment to the date of documented progression, or the date of death (in the absence of progression) of participants. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Pharmacokinetics (PK) parameter for total antibody (TAb): Maximum concentration (Cmax) | Dose 1 and Dose 3: pre-dose, 0.5 hour, 1 hour, 1.5 hours, 10 hours, 24 hours, 48 hours, 72 hours, 120 hours, 168 hours, 240 hours, 336 hours and 504 hours after start of infusion. Dose 2: pre-dose.
  Cmax will be derived from the PK blood samples collected.
PK parameter for TAb: Time to maximum concentration (Tmax) | Dose 1 and Dose 3: pre-dose, 0.5 hour, 1 hour, 1.5 hours, 10 hours, 24 hours, 48 hours, 72 hours, 120 hours, 168 hours, 240 hours, 336 hours and 504 hours after start of infusion. Dose 2: pre-dose.
  Tmax will be derived from the PK blood samples collected.
PK parameter for TAb: Area under the concentration-time curve (AUC) | Dose 1 and Dose 3: pre-dose, 0.5 hour, 1 hour, 1.5 hours, 10 hours, 24 hours, 48 hours, 72 hours, 120 hours, 168 hours, 240 hours, 336 hours and 504 hours after start of infusion. Dose 2: pre-dose.
  AUC will be derived from the PK blood samples collected.
PK parameter for TAb: Trough concentration (Ctrough) | Dose 1 and Dose 3: pre-dose, 0.5 hour, 1 hour, 1.5 hours, 10 hours, 24 hours, 48 hours, 72 hours, 120 hours, 168 hours, 240 hours, 336 hours and 504 hours after start of infusion. Dose 2: pre-dose.
  Ctrough will be derived from the PK blood samples collected.
PK parameter for TAb: Terminal or apparent terminal half-life (t1/2) | Dose 1 and Dose 3: pre-dose, 0.5 hour, 1 hour, 1.5 hours, 10 hours, 24 hours, 48 hours, 72 hours, 120 hours, 168 hours, 240 hours, 336 hours and 504 hours after start of infusion. Dose 2: pre-dose.
  t1/2 will be derived from the PK blood samples collected.
PK parameter for TAb: Systemic clearance (CL) | Dose 1 and Dose 3: pre-dose, 0.5 hour, 1 hour, 1.5 hours, 10 hours, 24 hours, 48 hours, 72 hours, 120 hours, 168 hours, 240 hours, 336 hours and 504 hours after start of infusion. Dose 2: pre-dose.
  CL will be derived from the PK blood samples collected.
PK parameter for antibody-drug conjugate (ADC): Cmax | Dose 1 and Dose 3: pre-dose, 0.5 hour, 1 hour, 1.5 hours, 10 hours, 24 hours, 48 hours, 72 hours, 120 hours, 168 hours, 240 hours, 336 hours and 504 hours after start of infusion. Dose 2: pre-dose.
  Cmax will be derived from the PK blood samples collected.
PK parameter for ADC: Tmax | Dose 1 and Dose 3: pre-dose, 0.5 hour, 1 hour, 1.5 hours, 10 hours, 24 hours, 48 hours, 72 hours, 120 hours, 168 hours, 240 hours, 336 hours and 504 hours after start of infusion. Dose 2: pre-dose.
  Tmax will be derived from the PK blood samples collected.
PK parameter for ADC: AUC | Dose 1 and Dose 3: pre-dose, 0.5 hour, 1 hour, 1.5 hours, 10 hours, 24 hours, 48 hours, 72 hours, 120 hours, 168 hours, 240 hours, 336 hours and 504 hours after start of infusion. Dose 2: pre-dose.
  AUC will be derived from the PK blood samples collected.
PK parameter for ADC: Ctrough | Dose 1 and Dose 3: pre-dose, 0.5 hour, 1 hour, 1.5 hours, 10 hours, 24 hours, 48 hours, 72 hours, 120 hours, 168 hours, 240 hours, 336 hours and 504 hours after start of infusion. Dose 2: pre-dose.
  Ctrough will be derived from the PK blood samples collected.
PK parameter for ADC: t1/2 | Dose 1 and Dose 3: pre-dose, 0.5 hour, 1 hour, 1.5 hours, 10 hours, 24 hours, 48 hours, 72 hours, 120 hours, 168 hours, 240 hours, 336 hours and 504 hours after start of infusion. Dose 2: pre-dose.
  t1/2 will be derived from the PK blood samples collected.
PK parameter for ADC: CL | Dose 1 and Dose 3: pre-dose, 0.5 hour, 1 hour, 1.5 hours, 10 hours, 24 hours, 48 hours, 72 hours, 120 hours, 168 hours, 240 hours, 336 hours and 504 hours after start of infusion. Dose 2: pre-dose.
  CL will be derived from the PK blood samples collected.
PK parameter for Monomethyl Auristatin E (MMAE): Cmax | Dose 1 and Dose 3: pre-dose, 0.5 hour, 1 hour, 1.5 hours, 10 hours, 24 hours, 48 hours, 72 hours, 120 hours, 168 hours, 240 hours, 336 hours and 504 hours after start of infusion. Dose 2: pre-dose.
  Cmax will be derived from the PK blood samples collected.
PK parameter for MMAE: Tmax | Dose 1 and Dose 3: pre-dose, 0.5 hour, 1 hour, 1.5 hours, 10 hours, 24 hours, 48 hours, 72 hours, 120 hours, 168 hours, 240 hours, 336 hours and 504 hours after start of infusion. Dose 2: pre-dose.
  Tmax will be derived from the PK blood samples collected.
PK parameter for MMAE: AUC | Dose 1 and Dose 3: pre-dose, 0.5 hour, 1 hour, 1.5 hours, 10 hours, 24 hours, 48 hours, 72 hours, 120 hours, 168 hours, 240 hours, 336 hours and 504 hours after start of infusion. Dose 2: pre-dose.
  AUC will be derived from the PK blood samples collected.
PK parameter for MMAE: Ctrough | Dose 1 and Dose 3: pre-dose, 0.5 hour, 1 hour, 1.5 hours, 10 hours, 24 hours, 48 hours, 72 hours, 120 hours, 168 hours, 240 hours, 336 hours and 504 hours after start of infusion. Dose 2: pre-dose.
  Ctrough will be derived from the PK blood samples collected.
PK parameter for MMAE: t1/2 | Dose 1 and Dose 3: pre-dose, 0.5 hour, 1 hour, 1.5 hours, 10 hours, 24 hours, 48 hours, 72 hours, 120 hours, 168 hours, 240 hours, 336 hours and 504 hours after start of infusion. Dose 2: pre-dose.
  t1/2 will be derived from the PK blood samples collected.
PK parameter for MMAE: CL | Dose 1 and Dose 3: pre-dose, 0.5 hour, 1 hour, 1.5 hours, 10 hours, 24 hours, 48 hours, 72 hours, 120 hours, 168 hours, 240 hours, 336 hours and 504 hours after start of infusion. Dose 2: pre-dose.
  CL will be derived from the PK blood samples collected.
Immunogenicity assessment | Dose 1 to Dose 3: pre-dose, and 504 hours after start of infusion (Dose 3 only)
  Assessment of anti-RC108 antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Yuankai Shi, M.D., Principal Investigator — Cancer Hospital, Chinese Academy of Medical Science and Peking Union Medical College
Locations (4):
- China (4):
  - National Cancer Center/Cancer Hospital, Chinese Academy of Medical Science and Peking Union Medical College, Beijing, Beijing Municipality
  - Hunan Cancer Hospital, Changsha, Hunan
  - The First Hospital of Jilin University, Changchun, Jilin
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No